CLINICAL TRIAL: NCT00267007
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, 18 Week Pilot Study to Investigate the Neuroprotective Effect of PROCRIT (Epoetin Alfa) on the Development of Peripheral Neuropathy in Patients Receiving Combination Taxane and Platinum-Based Chemotherapy for Cancer
Brief Title: A Study to Investigate the Neuroprotective Effect of PROCRIT (Epoetin Alfa) Versus Placebo in Cancer Patients Who Develop Chemotherapy-induced Peripheral Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CR003247
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Results first posted 2009-09-07 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Peripheral Neuropathy, Chemotherapy-induced
Keywords: Peripheral neuropathy; Chemotherapy-induced; Hemoglobin level; Cancer; Taxane; Platinum-based chemotherapy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neoplasms | interventions — Epoetin Alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 (Experimental): PROCRIT 40 000 IU QW Epoetin alpha (PROCRIT) 40 000 IU every week (QW) for 18 weeks (IV or SC)
  Interventions: Drug: PROCRIT 40,000 IU QW
- 002 (Placebo Comparator): Placebo Equivalent volume to PROCRIT (1 mL) administered (QW) for 18 weeks (IV or SC)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PROCRIT 40,000 IU QW — Epoetin alpha (PROCRIT) 40,000 IU every week (QW) for 18 weeks (IV or SC)
  Arms: 001
Drug: Placebo — Equivalent volume to PROCRIT (1 mL) administered (QW) for 18 weeks (IV or SC)
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the neuroprotective effect of PROCRIT (epoetin alfa, a glycoprotein that stimulates red blood cell production) versus placebo in patients with cancer who develop chemotherapy-induced peripheral neuropathy due to combination Taxane and Platinum-Based treatment.

DETAILED DESCRIPTION:
Peripheral neuropathy is a debilitating disease of the nerves which can be a dose-limiting toxicity of chemotherapeutic agents. The symptoms of peripheral neuropathy can lead to considerable patient distress and discomfort, discontinuation of chemotherapy, and limitations regarding the selection of future chemotherapeutic regimens. Symptoms such as numbness, weakness, burning pain (especially at night), and loss of reflexes may take months before they improve and permanent deficits may remain. Epoetin alfa, already used in the treatment of chemotherapy-induced anemia, has been shown to have neuroprotective effects in preclinical studies. The purpose of this randomized (patients are assigned different treatments based on chance), double-blind (neither the patient nor the physician knows whether drug or placebo is being taken, or at what dosage), placebo-controlled study is to evaluate the neuroprotective effect of PROCRIT (epoetin alfa) administered once every week in patients with cancer who develop chemotherapy-induced peripheral neuropathy due to treatment with combination Taxane and Platinum-Based chemotherapy. Patients will receive injections subcutaneously or intravenously of either epoetin alfa or placebo once weekly for up to 18 weeks. Doses may be adjusted in the range of 20,000 to 60,000 Units once a week, depending on the patient's hemoglobin levels. Safety evaluations will be conducted throughout the study at specified intervals and will consist of assessment of laboratory tests (Hemoglobin level, Complete Blood Count (CBC), Blood Chemistries), vital signs, physical examinations and occurrence and severity of adverse events. In addition, the occurrence of anti-erythropoietin antibodies at baseline and study completion/early withdrawal will be evaluated in patients who received PROCRIT (Epoetin alfa) after database lock and unblinding has occurred. The primary measure of effectiveness is the change at Week 12 in the National Cancer Institute Common Toxicity Criteria (NCI CTC) neuropathy score. The study hypothesis is that epoetin alfa will be more effective in the treatment of chemotherapy-induced peripheral neuropathy than placebo as measured at Week 12 by the National Cancer Institute Common Toxicity Criteria (NCI CTC) neuropathy score. Patients will receive injections subcutaneously (SC, under the skin) or intravenously (IV, in a vein) of either epoetin alfa or placebo once weekly for up to 18 weeks. Doses may be adjusted depending on the patient's hemoglobin levels to the maximum 60,000 Units once a week. The minimum dose can be 20,000 Units once a week.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of cancer , and no history of peripheral neuropathy
* Have had the appropriate surgery for carcinoma and are no more than 12 weeks post-operatively at study entry
* Have not received chemotherapy (chemotherapy naïve patients) and are scheduled to receive at least 4 cycles of combination taxane and platinum-based chemotherapy
* Have a hemoglobin value of >= 10 and < 12 g/dL
* have a life expectancy of at least 6 months

Exclusion Criteria:

* Patients who have had prior treatment with PROCRIT (epoetin alfa) or similar drugs (erythropoietic agents) within the last 2 months
* Have used experimental treatments within the last year that are reported or hypothesized to have neuroprotective potential, including amifostine, cyanocobalamin (vitamin B12), alpha-tocopherol (Vitamin E), glutamine, and gabapentin
* have anemia due to factors other than cancer/chemotherapy, or have ongoing neuropathy due to any cause
* Received a transfusion of platelets or packed red blood cells within 28 days prior to the first dose of study medication
* Have a history of pulmonary emboli, deep vein thrombosis, ischemic stroke or any other history of arterial or venous thrombotic events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (28):
- United States (28):
  - Mobile, Alabama
  - Little Rock, Arkansas
  - Alhambra, California
  - Bakersfield, California
  - Fullerton, California
  - La Verne, California
  - Long Beach, California
  - Northridge, California
  - Oxnard, California
  - Santa Maria, California
  - New Haven, Connecticut
  - Hollywood, Florida
  - Augusta, Georgia
  - Joliet, Illinois
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Bethesda, Maryland
  - Detroit, Michigan
  - Southfield, Michigan
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Buffalo, New York
  - Syracuse, New York
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Chattanooga, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- PROCRIT 40,000 IU QW: Epoetin alpha (PROCRIT) 40,000 IU every week (QW) for 18 weeks (intravenous or subcutaneous)
- Placebo: Equivalent volume to PROCRIT (1 mL) administered every week (QW) for 18 weeks (intravenous or subcutaneous)
Period: Overall Study
Arm/Group | PROCRIT 40,000 IU QW | Placebo
Started | 19 (2 additional patients were randomized but never received study medication and no data were collected) | 11
Completed | 11 | 10
Not Completed | 8 | 1
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Non-compliance | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PROCRIT 40,000 IU QW | Placebo | Total
Number analyzed (Participants) | 19 | 11 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 8 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (14.18) | 56.8 (12.98) | 58.9 (13.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 11 | 30
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Developed Peripheral Sensory Neuropathy (National Cancer Institute Common Toxicity Criteria (NCI CTC) Score >= 1) at Week 12.
Description: NCI CTC neuropathy: a descriptive terminology used to grade the severity of AEs in cancer subjects on a 0-5 scale. A higher score indicates worse peripheral neuropathy.
Time Frame: Baseline to Week 12
Population: MITT(Modified intent to treat)all randomized subjects that received at least one dose and had at least one post-baseline neuropathy assessment.
Measure: Number; unit: participants
Arm/Group | PROCRIT 40,000 IU QW | Placebo
Number analyzed (Participants) | 19 | 11
participants | 5 | 6

2. Secondary Outcome: The Number of Patients Who Developed Peripheral Sensory Neuropathy (National Cancer Institute Common Toxicity Criteria (NCI CTC) Score >= 2) at Week 12.
Description: as for outcome 1
Time Frame: baseline to Day 128
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | PROCRIT 40,000 IU QW | Placebo
Number analyzed (Participants) | 19 | 11
participants | 3 | 0

ADVERSE EVENTS:
Arm/Group | PROCRIT 40,000 IU QW | Placebo
Serious Adverse Events (participants affected / at risk) | 6 | 1
Other Adverse Events (participants affected / at risk) | 19 | 11
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | PROCRIT 40,000 IU QW | Placebo
Intestinal Obstruction (Gastrointestinal disorders) | 1/19 | 0/11
Small Intestinal Obstruction (Gastrointestinal disorders) | 1/19 | 1/11
Post Procedural Cellulitis (Infections and infestations) | 1/19 | 0/11
Dehydration (Metabolism and nutrition disorders) | 1/19 | 0/11
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/19 | 0/11
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1/19 | 0/11
Lymphocele (Vascular disorders) | 1/19 | 0/11
Thrombophlebitis Superficial (Vascular disorders) | 1/19 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | PROCRIT 40,000 IU QW | Placebo
Anaemia (Blood and lymphatic system disorders) | 3/19 | 2/11
Bone Marrow Failure (Blood and lymphatic system disorders) | 0/19 | 1/11
Leukopenia (Blood and lymphatic system disorders) | 1/19 | 0/11
Neutropenia (Blood and lymphatic system disorders) | 7/19 | 4/11
Thrombocytopenia (Blood and lymphatic system disorders) | 6/19 | 2/11
Tachycardia (Cardiac disorders) | 1/19 | 0/11
Diplopia (Eye disorders) | 1/19 | 0/11
Dry Eye (Eye disorders) | 0/19 | 1/11
Lacrimation Increased (Eye disorders) | 1/19 | 0/11
Vision Blurred (Eye disorders) | 1/19 | 1/11
Abdominal Pain (Gastrointestinal disorders) | 5/19 | 2/11
Abdominal Pain Upper (Gastrointestinal disorders) | 1/19 | 0/11
Anal Discomfort (Gastrointestinal disorders) | 1/19 | 0/11
Constipation (Gastrointestinal disorders) | 9/19 | 5/11
Diarrhoea (Gastrointestinal disorders) | 3/19 | 4/11
Flatulence (Gastrointestinal disorders) | 1/19 | 1/11
Haemorrhoids (Gastrointestinal disorders) | 0/19 | 1/11
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1/19 | 0/11
Nausea (Gastrointestinal disorders) | 16/19 | 8/11
Odynophagia (Gastrointestinal disorders) | 2/19 | 0/11
Small Intestinal Obstruction (Gastrointestinal disorders) | 1/19 | 0/11
Stomatitis (Gastrointestinal disorders) | 3/19 | 2/11
Toothache (Gastrointestinal disorders) | 1/19 | 0/11
Vomiting (Gastrointestinal disorders) | 8/19 | 7/11
Asthenia (General disorders) | 4/19 | 2/11
Catheter Site Erythema (General disorders) | 0/19 | 1/11
Catheter Site Pain (General disorders) | 0/19 | 2/11
Fatigue (General disorders) | 16/19 | 8/11
Injection Site Reaction (General disorders) | 1/19 | 0/11
Mucosal Inflammation (General disorders) | 2/19 | 3/11
Non-Cardiac Chest Pain (General disorders) | 2/19 | 0/11
Oedema (General disorders) | 2/19 | 0/11
Odema Peripheral (General disorders) | 0/19 | 1/11
Pain (General disorders) | 1/19 | 0/11
Pyrexia (General disorders) | 5/19 | 0/11
Drug Hypersensitivity (Immune system disorders) | 1/19 | 0/11
Catheter Site Infection (Infections and infestations) | 1/19 | 1/11
Fungal Infection (Infections and infestations) | 2/19 | 0/11
Gastroenteritis (Infections and infestations) | 0/19 | 1/11
Herpes Simplex (Infections and infestations) | 1/19 | 0/11
Pneumonia (Infections and infestations) | 1/19 | 0/11
Post Procedural Infection (Infections and infestations) | 1/19 | 0/11
Respiratory Tract Infection (Infections and infestations) | 0/19 | 1/11
Rhinitis (Infections and infestations) | 3/19 | 2/11
Sinusitis (Infections and infestations) | 1/19 | 0/11
Upper Respiratory Tract Infection (Infections and infestations) | 2/19 | 0/11
Urinary Tract Infection (Infections and infestations) | 2/19 | 0/11
Vaginal Infection (Infections and infestations) | 1/19 | 0/11
Viral Infection (Infections and infestations) | 1/19 | 0/11
Vulvovaginal Mycotic Infection (Infections and infestations) | 1/19 | 0/11
Contusion (Injury, poisoning and procedural complications) | 1/19 | 1/11
Excoriation (Injury, poisoning and procedural complications) | 1/19 | 1/11
Feeding Tube Complication (Injury, poisoning and procedural complications) | 0/19 | 1/11
Incision Site Complication (Injury, poisoning and procedural complications) | 1/19 | 0/11
Incision Site Pain (Injury, poisoning and procedural complications) | 1/19 | 1/11
Joint Sprain (Injury, poisoning and procedural complications) | 0/19 | 1/11
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0/19 | 1/11
Procedural Pain (Injury, poisoning and procedural complications) | 1/19 | 0/11
Procedural Site Reaction (Injury, poisoning and procedural complications) | 1/19 | 0/11
Blood Alkaline Phosphatase Increased (Investigations) | 1/19 | 0/11
Blood Calcium Decreased (Investigations) | 1/19 | 0/11
Blood Magnesium Decreased (Investigations) | 1/19 | 0/11
Electrocardiogram QT Prolonged (Investigations) | 1/19 | 0/11
Haemoglobin Decreased (Investigations) | 2/19 | 0/11
Heart Rate Increased (Investigations) | 1/19 | 0/11
Neutrophil Count Decreased (Investigations) | 0/19 | 1/11
Urine Output Decreased (Investigations) | 1/19 | 0/11
White Blood Cell Count Decreased (Investigations) | 1/19 | 0/11
Anorexia (Metabolism and nutrition disorders) | 6/19 | 3/11
Dehydration (Metabolism and nutrition disorders) | 0/19 | 1/11
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0/19 | 1/11
Hyperglycaemia (Metabolism and nutrition disorders) | 1/19 | 0/11
Hyperkalaemia (Metabolism and nutrition disorders) | 1/19 | 0/11
Hypocalcaemia (Metabolism and nutrition disorders) | 2/19 | 0/11
Hypochloraemia (Metabolism and nutrition disorders) | 1/19 | 0/11
Hypokalaemia (Metabolism and nutrition disorders) | 4/19 | 1/11
Hypomagnesaemia (Metabolism and nutrition disorders) | 4/19 | 1/11
Hyponatraemia (Metabolism and nutrition disorders) | 2/19 | 0/11
Arthralgia (Musculoskeletal and connective tissue disorders) | 9/19 | 4/11
Back Pain (Musculoskeletal and connective tissue disorders) | 1/19 | 2/11
Bone Pain (Musculoskeletal and connective tissue disorders) | 1/19 | 0/11
Groin Pain (Musculoskeletal and connective tissue disorders) | 1/19 | 0/11
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1/19 | 0/11
Lower Extremity Mass (Musculoskeletal and connective tissue disorders) | 0/19 | 1/11
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3/19 | 0/11
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 0/19 | 2/11
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0/19 | 1/11
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1/19 | 1/11
Myalgia (Musculoskeletal and connective tissue disorders) | 7/19 | 4/11
Neck Pain (Musculoskeletal and connective tissue disorders) | 0/19 | 1/11
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3/19 | 1/11
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/19 | 0/11
Dizziness (Nervous system disorders) | 2/19 | 2/11
Dysgeusia (Nervous system disorders) | 4/19 | 1/11
Headache (Nervous system disorders) | 4/19 | 4/11
Hypoaesthesia (Nervous system disorders) | 4/19 | 1/11
Paraesthesia (Nervous system disorders) | 3/19 | 3/11
Perripheral Motor Neuropathy (Nervous system disorders) | 6/19 | 3/11
Peripheral Sensory Neuropathy (Nervous system disorders) | 11/19 | 9/11
Syncope (Nervous system disorders) | 0/19 | 2/11
Anxiety (Psychiatric disorders) | 1/19 | 1/11
Confusional State (Psychiatric disorders) | 1/19 | 0/11
Depression (Psychiatric disorders) | 0/19 | 1/11
Insomia (Psychiatric disorders) | 7/19 | 1/11
Mood Altered (Psychiatric disorders) | 1/19 | 0/11
Sleep Disorder (Psychiatric disorders) | 1/19 | 0/11
Bladder Spasm (Renal and urinary disorders) | 1/19 | 0/11
Dysuria (Renal and urinary disorders) | 2/19 | 0/11
Haematuria (Renal and urinary disorders) | 0/19 | 1/11
Proteinuria (Renal and urinary disorders) | 0/19 | 1/11
Menopausal Symptons (Reproductive system and breast disorders) | 1/19 | 0/11
Pelvic Pain (Reproductive system and breast disorders) | 1/19 | 0/11
Vaginal Discharge (Reproductive system and breast disorders) | 1/19 | 1/11
Vaginal Ulceration (Reproductive system and breast disorders) | 0/19 | 1/11
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1/19 | 0/11
Cough (Respiratory, thoracic and mediastinal disorders) | 4/19 | 2/11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3/19 | 2/11
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 2/19 | 1/11
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1/19 | 0/11
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0/19 | 1/11
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1/19 | 0/11
Alopecia (Skin and subcutaneous tissue disorders) | 10/19 | 5/11
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1/19 | 0/11
Dry Skin (Skin and subcutaneous tissue disorders) | 1/19 | 0/11
Nail Disorder (Skin and subcutaneous tissue disorders) | 1/19 | 0/11
Petechiae (Skin and subcutaneous tissue disorders) | 0/19 | 1/11
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1/19 | 0/11
Pruritus (Skin and subcutaneous tissue disorders) | 0/19 | 1/11
Rash (Skin and subcutaneous tissue disorders) | 3/19 | 2/11
Rash Macular (Skin and subcutaneous tissue disorders) | 0/19 | 1/11
Flushing (Vascular disorders) | 2/19 | 1/11
Hot Flush (Vascular disorders) | 2/19 | 1/11
Hypertension (Vascular disorders) | 1/19 | 0/11
Hypotension (Vascular disorders) | 2/19 | 0/11
Lymphocele (Vascular disorders) | 1/19 | 0/11
Lymphoedema (Vascular disorders) | 1/19 | 0/11
Dry Mouth (Gastrointestinal disorders) | 0/19 | 1/11
Dyspepsia (Gastrointestinal disorders) | 5/19 | 2/11
Dysphagia (Gastrointestinal disorders) | 1/19 | 0/11

LIMITATIONS AND CAVEATS:
No formal analysis was conducted due to early termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less